CLINICAL TRIAL: NCT06504368
Title: An Open-Label, Phase 1, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous DCR-PDL1 in Adults With Solid Tumors
Brief Title: Safety, Tolerability, and Pharmacokinetics of DCR-PDL1 in Adults With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCR-PDL1-101
Record Dates: First submitted 2024-06-18; First posted 2024-07-16 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DCR-PDL1 (Experimental): Participants will receive multiple IV doses of DCR-PDL1 during each treatment cycle.
  Interventions: Drug: DCR-PDL1

INTERVENTIONS:
Drug: DCR-PDL1 — Solution for IV Infusion

SUMMARY:
The study will evaluate the safety, tolerability, and pharmacokinetics of intravenous DCR-PDL1 in adults with solid tumors. Participants will be enrolled in one of 4 ascending-dose cohorts. Each treatment cycle will consist of multiple intravenous (IV) doses. Dose escalation decisions will be based on data collected during the dose-limiting toxicity (DLT) period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, aged greater than or equal to (≥) 18 years.
* Participants are required to have a documented, locally advanced or metastatic solid tumor malignancy, or non-Hodgkin's lymphoma

  * that is refractory to standard therapy known to provide clinical benefit for their condition OR
  * have demonstrated evidence of disease progression or relapse, via imaging, during or following standard therapy known to provide clinical benefit for their condition, OR
  * have demonstrated intolerance to standard therapy known to provide clinical benefit for their condition. OR
  * for which no standard therapy is available
* Measurable disease according to RECIST version 1.1.
* Malignancy not currently amenable to surgical intervention.
* ECOG performance status of 0, 1, or 2, and an anticipated life expectancy of ≥ 3 months at the time of signing the informed consent.
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with known CNS or leptomeningeal metastases not controlled by prior surgery or radiotherapy, or symptoms suggesting CNS involvement for which treatment is required.
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Nature of Adverse Events (AEs) | Baseline to week 8
Incidence of Dose-limiting Toxicities (DLTs) | Baseline to week 8
Change From Baseline in Vital Signs: Oral, Tympanic, Temporal Artery Temperature | Baseline up to week 8
  Vital signs will be measured in a semi-supine (i.e., semi-recumbent) position.
Change From Baseline in Vital Signs: Systolic and Diastolic Blood Pressure | Baseline up to week 8
  Vital signs will be measured in a semi-supine (i.e., semi-recumbent) position.
Change From Baseline in Vital Signs: Pulse and Respiratory Rate | Baseline up to week 8
  Vital signs will be measured in a semi-supine (i.e., semi-recumbent) position. Blood pressure and pulse measurements should be preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Change from Baseline in 12-lead Electrocardiogram (ECG): Heart Rate and Pulse Rate | Baseline to week 8
Change from Baseline in 12-lead Electrocardiogram (ECG): QRS intervals | Baseline to week 8
  ECG recordings will be made in a semi-supine (i.e., semi-recumbent) position, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Change from Baseline in 12-lead Electrocardiogram (ECG): QT intervals | Baseline to week 8
  ECG recordings will be made in a semi-supine (i.e., semi-recumbent) position, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Change from Baseline in 12-lead Electrocardiogram (ECG): QTcF intervals (QT Interval Corrected by the Fridericia Formula) | Baseline to week 8
  ECG recordings will be made in a semi-supine (i.e., semi-recumbent) position, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Change from Baseline in Hematology Parameter: Red blood cells, White blood cells, Lymphocytes, Monocytes, Eosinophils, Neutrophils, Basophils and Platelets, Reticulocytes | Baseline to week 8
Change from Baseline in Hematology Parameter: Mean corpuscular volume (MCV) | Baseline to week 8
Change from Baseline in Hematology Parameter: Mean corpuscular hemoglobin (MCH) | Baseline to week 8
Change from Baseline in Hematology Parameter: Hemoglobin | Baseline to week 8
Change from Baseline in Hematology Parameter: Hematocrit and Mean corpuscular hemoglobin concentration (MCHC) | Baseline to week 8
Change from Baseline in Coagulation Parameter: International normalized ratio (INR) | Baseline to week 8
Change from Baseline in Coagulation Parameter: Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) | Baseline to week 8
Change from Baseline in Coagulation Parameter: Fibrinogen | Baseline to week 8
Change from Baseline in Clinical Chemistry Parameter: Alanine transaminase (ALT), Aspartate transaminase (AST), Gamma-glutamyl transferase (GGT), Alkaline phosphatase (ALP), Lactate dehydrogenase (LDH) and Creatine kinase (CK) | Baseline to week 8
Change from Baseline in Clinical Chemistry Parameter: Total protein and Albumin | Baseline to week 8
Change from Baseline in Clinical Chemistry Parameter: Total bilirubin, Direct bilirubin, Fasting blood glucose, Creatinine and Blood urea nitrogen (BUN) | Baseline to week 8
Change from Baseline in Clinical Chemistry Parameter: Sodium, Chloride and Potassium | Baseline to week 8
Change from Baseline in Urinalysis Parameter: Glucose, Protein, Bilirubin and Urobilinogen | Baseline to week 8
Change from Baseline in Urinalysis Parameter: Specific Gravity | Baseline to week 8
Change from Baseline in Urinalysis Parameter: Potential of Hydrogen (pH) of Urine | Baseline to week 8
Change from Baseline in Urinalysis Parameter: Blood | Baseline to week 8
Change from Baseline in Urinalysis Parameter: Ketones and Nitrite | Baseline to week 8
Change from Baseline in Urinalysis Parameter: Leukocyte esterase | Baseline to week 8
Number of Participants with Change from Baseline in Physical Examination Findings: Cardiovascular, Respiratory, Gastrointestinal, and Neurological systems | Baseline to week 8
  A complete physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal, and neurological systems.

SECONDARY OUTCOMES:
Pharmacokinetic Plasma Concentrations of DCR-PDL1 | Pre-dose up to 48 hours post-dose
Pharmacokinetic Urine Concentrations of DCR-PDL1 | Up to 8 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - NEXT Oncology, Irving, Texas
  - Next Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No